CLINICAL TRIAL: NCT05469373
Title: Electrical Stimulation for Seizure Induction in Pediatric Drug-Refractory Epilepsy (ESIS in Pedriatric DRE).
Brief Title: ESIS in Pediatric DRE
Status: Recruiting | Type: Observational
Sponsor: Sarah Katie Ihnen (Other)
Collaborators: Network for Excellence in Neuroscience Clinical Trials (Unknown); Child Neurologist Career Development Program (Unknown)
Responsible Party: Sponsor-Investigator, Sarah Katie Ihnen, Faculty, Research Instructor, Children's Hospital Medical Center, Cincinnati
Organization: Children's Hospital Medical Center, Cincinnati (Other)
Other Study IDs: 2022-0020
Record Dates: First submitted 2022-06-23; First posted 2022-07-21 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Epilepsy
Keywords: epilepsy surgery, drug-resistant epilepsy, tuberous sclerosis
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy; Tuberous Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main reason for this research study is to gain information about how the brain makes seizures by causing seizures using very small amounts of current, or electrical stimulation. Using small amounts of current to cause seizures (or stimulate) is not new at CCHMC - it is part of routine clinical practice for some patients at some electrodes.

This study differs from routine clinical care in that all study patients will undergo electrical stimulation in all or nearly all electrode contacts. The study team is doing this because there is promising data in adult patients that stimulating comprehensively (targeting all or nearly all of the electrode contacts) helps define the seizure network. Defining the seizure network in turn helps the medical team plan surgery. So far, there is not as much published data on seizure stimulation for pediatric patients.

This research study thus has the potential both to help individual patients (by providing specific information about your seizure networks) and to help pediatric patients with epilepsy in general (by increasing our understanding of stimulated seizures in children, teenagers and young adults).

DETAILED DESCRIPTION:
Epilepsy affects about 1% of the population, with roughly 30% of patients with epilepsy eventually developing drug-resistant epilepsy (DRE). Increasingly, surgery is pursued for DRE, yielding seizure freedom rates of 50-70%. However, accurate deduction of the epileptogenic zone (EZ) for surgical planning can be difficult in pediatric DRE, especially in those cases of multifocal seizures, as is often seen in Tuberous Sclerosis Complex (TSC), for example. Patients with multifocal epilepsy typically require a period of pre-surgical invasive EEG monitoring to record spontaneous seizures, the gold standard for EZ deduction. Unfortunately, the invasive monitoring process may be lengthy, costly and even fail to reveal a dominant EZ.

Electrical stimulation of induced seizures (ESIS) using stereo EEG (sEEG) has been shown to be a safe and valid adjunct for EZ delineation in adults with DRE. ESIS can be implemented within 1-2 days of electrode implantation, while the patient would otherwise be passively awaiting spontaneous seizures. ESIS typically induces habitual seizures with few side effects, and there is no data to suggest that ESIS inhibits spontaneous seizures or prolongs the otherwise clinically-indicated hospital stay. Crucially, published data show that induced seizures provide information about the EZ that is both convergent with and unique from that provided by spontaneous seizures. Despite these promising reports, ESIS is not widely integrated into pediatric DRE evaluation.

The overall objective is to improve methods of EZ identification in pediatric DRE patients with complex EZs, thereby increasing the likelihood of surgical candidacy for patients and ultimately improving surgical outcomes. In this protocol, investigators hypothesize that electrical stimulation of induced seizures (ESIS) is an effective adjunct for EZ delineation in children with DRE. To test this, the study will enroll n=86 patients with DRE undergoing sEEG evaluation aged 1-30 years. Based on the CCHMC epilepsy surgery program throughput, it is anticipated that this will include approximately n=36 patients with TSC and n=50 without TSC, which will provide the opportunity to compare the utility of this technique between patients with and without TSC. Patients will undergo ESIS using published Cincinnati Children's Hospital Medical Center (CCHMC) parameters with modifications. Gray and white matter contacts will be stimulated systematically. Safety, tolerability, yield, validity and parameter space will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of drug-refractory epilepsy (DRE)
* 1-30 years of age
* recommended to undergo stereoencephalography (sEEG) at CCHMC

Exclusion Criteria:

* <1 and >30 years of age

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants with drug-refractory epilepsy who receive care at or are referred into the CCHMC Comprehensive Epilepsy Center will comprise the targeted study population. Specifically, those patients who undergo phase I evaluations and are subsequently recommended for phase II evaluations at CCHMC will be identified as research study candidates.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety -- Occurrence of generalized, convulsive and prolonged seizures | Phase II epilepsy surgery testing
  Evaluate the safety of ESIS in pediatric DRE patients.
Tolerability -- Quantify study withdrawal and patient/caregiver experience | during Phase II epilepsy surgery testing
  Evaluate the tolerability of ESIS in pediatric DRE patients.
Yield -- Rate of induction of habitual seizures | during Phase II epilepsy surgery testing
  Evaluate the yield of ESIS in pediatric DRE patients.
Clinical Validity | during Phase II epilepsy surgery testing and through study completion, an average of 1 year
  Test the clinical validity of ESIS in pediatric DRE patients by examining the impact of occurance of induced seizures on surgical outcomes.
Predictors | during Phase II epilepsy surgery testing
  Investigate the methodologic, anatomic, and patient-specific predictors of induced seizures in pediatric DRE patients.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Katie Ihnen, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States